CLINICAL TRIAL: NCT04154163
Title: Appropriate Dosing to Optimise Personalised Cancer Treatments
Acronym: ADOPT
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: 2-032-19
Record Dates: First submitted 2019-10-31; First posted 2019-11-06 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Melanoma Stage III; Melanoma Stage IV; Ovarian Cancer; Renal Cancer Stage III; Renal Cancer Stage IV; Lung Cancer, Non-small Cell
MeSH Terms: conditions — Melanoma; Ovarian Neoplasms; Kidney Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Dried Blood Spot Testing; Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimens will be blood tests conducted in the form of either (i) whole blood which will be collected using Dried Blood Spots "DBS" +/- and (ii) venous blood samples.
  Stage 1:
  Five patients will be recruited for initial validation of drug dose measurements using the DBS method by comparison with venous blood samples.
  One or two drops of blood (10 microlitres) collected using triplicates of blood spots on to dry blood spot filter paper and micro-sampler sponge at specified time intervals.
  A phlebotomy serum sample (5 ml) will be collected in a heparin tube at the same time intervals before and after oral dosing of their targeted drugs over a single 24-hour period.
  Stage 2:
  One or two drops of blood (10 microlitres) collected using triplicates of blood spots on to dry blood spot filter paper and micro-sampler sponge at specified time intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1 Participants: Blood test Day 1 DBS and venous blood
  Blood test Day 2 DBS (+/- and venous blood)
  Blood test Day 15 DBS only
  Blood test Day 16 DBS only
  Interventions: Diagnostic Test: Dried blood Spot (DBS); Diagnostic Test: Venous blood sampling
- Stage 2 Participants: Non-drug naive participants:
  Blood test Day 1 DBS
  Blood test Day 2 DBS
  Blood test Day 15 DBS
  Blood test Day 16 DBS
  Drug naive participants:
  Blood test Day 1 DBS
  Blood test Day 2 DBS
  Blood test Day 3, 4, or 5 DBS
  Blood test Day 4, 5 or 6 DBS
  Blood test Day 15 DBS
  Blood test Day 16 DBS
  Interventions: Diagnostic Test: Dried blood Spot (DBS)

INTERVENTIONS:
Diagnostic Test: Dried blood Spot (DBS) — Dried Blood Spot filter paper and sponges
  Other Names: DBS home collection kits
Diagnostic Test: Venous blood sampling — Venous blood
  Other Names: Phlebotomy
  Groups: Stage 1 Participants

SUMMARY:
This is a pilot study to assess feasibility of dried blood spot (DBS) samples for pharmacokinetic measurements of targeted anti-cancer drugs in oncology patients such as patients with BRAF-mutant melanoma receiving targeted treatment with BRAF and MEK inhibitors.

DETAILED DESCRIPTION:
In the pharmacology laboratory, we have developed a method for measuring drug concentrations in animals using dried blood spots (DBS). DBS is a simple method that could be easily carried out by patients at home, using either filter paper-based DBS cards (e.g. Whatman 903, FTA DMPK-C) or small sponges (www.neoteryx.com).

The routine use of DBS to clinically test blood was first used in the 1960s as a safe and simple method of testing for inherited metabolic disorders in new born babies. However, in recent years there has been increasing use of DBS to test blood for other things, including for drugs as a way to monitor the drug level in the blood.

This method has great potential application in testing blood for drug levels in cancer patients. We wish to establish if this DBS technique is feasible in real-life practice for cancer patients on targeted anti-cancer therapies as should this be the case this innovation could herald a new era in personalised treatment of advanced human cancers allowing doctors to more safely use combinations of targeted therapies. These combinations of targeted therapies have been shown to inhibit development of drug resistance and are increasingly being used in clinical practice. However, targeted therapies often fail (especially combinations of targeted therapies) because of unacceptable toxicities making them intolerable for the patient. With an easy and acceptable method for monitoring the drug level in blood, as could be provided by DBS, the right amount of drug could be given to each individual patient and this 'personalised' drug dosing as standard of care might result in much greater success with combinations of anti-cancer drugs.

This drug monitoring is especially important for targeted anti-cancer therapies because many of these (such as Dabrafenib, used for many cases of advanced melanoma) have profound affects on the liver enzymes that metabolise (get rid of) most medications. Dabrafenib is a potent inducer of P450 liver enzymes and this induction means that other drugs metabolised by the same liver pathway (the great majority of drugs are metabolised by the same pathways) will have significantly reduced blood levels if the patient is on Dabrafenib. So it is especially important to be able to monitor blood levels of both Dabrafenib and of other co-medications that the patient may be taking. The DBS sampling method would allow this and would provide a safe, convenient and cheap test that could be conducted in the patient's home and posted back to the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants
* Age 18 years and over
* Confirmed diagnosis of stage 4 or stage 3 unresectable cancers; BRAF+ melanoma, c-KIT+ melanoma, advanced renal cell carcinoma, non-small cell lung carcinoma and ovarian carcinoma.
* Able to perform study assessments
* Individuals who are participating in the follow-up phase of another interventional trial/study, or who are enrolled in an observational study, will be co-enrolled where the CIs of each study agree that it is appropriate

Exclusion Criteria:

* Inability to give informed consent
* World Health Organisation (WHO) performance status 3-4
* Known allergy or intolerance to Dabrafenib +/- Trametinib, Prazopanib, Erlotinib, Gefitinib, Imatinib, Osimertinib or Olaparib
* Unstable co-morbidities; cardiovascular disease e.g. severe congestive cardiac failure, end stage renal failure, hepatic impairment, vasculopathy, inflammatory arthritis or interstitial lung disease/ pneumonitis which, in the opinion of the CI, would make the patient unsuitable to be enrolled in the study
* Language barrier preventing adequate understanding of the study and a lack of suitable translator service to overcome this barrier
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Oncology Unit and Dermatology or Oncology outpatient departments
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
The accuracy of DBS for measuring drug levels in venous blood following standard doses of targeted therapies for metastatic cancers such as BRAF mutant melanoma | Pre-dose,1 hour, 2 hours, 8 hours (if on a once daily drug regime) or pre-second dose (if on a twice daily drug regime) and 24 hours post-dosing
  Concentration of targeted anti-cancer drug in venous blood at timed intervals following oral dosing in standard clinical care pathway measured in venous blood and by DBS

SECONDARY OUTCOMES:
The ability of oncology patients receiving targeted cancer treatments to collect multiple DBS samples over a 24-hour period | Pre-dose,1 hour, 2 hours, 8 hours (if on a once daily drug regime) or pre-second dose (if on a twice daily drug regime) and 24 hours post-dosing
  Successful collection of DBS samples both under supervision in hospital and when at home
The safety and acceptability of DBS collections at timed intervals before and after taking anti-cancer targeted drugs | After each 24-hour period of DBS sampling and during telephone consultations in weeks 1 and 4
  Number of Adverse Events per participant and measures of patient acceptability for collection of DBS
The stability of the drug levels stored in DBS, taken by the patient at home and posted to the laboratory | Measurement of repeat samples at the timepoints chosen at 1, 2 and 3-days post-collection to ensure stability.
  Demonstration that the drug concentrations measured in fresh and DBS samples stored for several days is the same.
Examine inter-patient variability in Pharmacokinetics (PK) | Measurement of co-medication drug levels at repeat time intervals (Pre-dose,1-hour, 2-hours, 8-hours (once-daily drug regime) or pre-second dose (twice-daily drug regime) and 24-hours post-dosing both before and after starting targeted Dabrafenib
  Changes in drug levels of co-medications over time following standard clinical dosing with targeted cancer treatments such as dabrafenib +/- trametinib
Drug tolerability collected from examination of clinical pathway for participating patients | Before recruitment and after commencing relevant medication
  Collection of drug tolerability data from examination of clinical pathway for participating patients

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Proby, MBBS,FRCP, Principal Investigator — Chief Investigator
Locations (1):
- NHS Tayside and University of Dundee, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
De-identified individual participants data for full primary and secondary outcome measures maybe be made available

REFERENCES:
- [Background] Robijns K, Koster RA, Touw DJ. Therapeutic drug monitoring by dried blood spot: progress to date and future directions. Clin Pharmacokinet. 2014 Nov;53(11):1053. doi: 10.1007/s40262-014-0197-3. No abstract available. PMID 25312497
- [Background] de Wit D, den Hartigh J, Gelderblom H, Qian Y, den Hollander M, Verheul H, Guchelaar HJ, van Erp NP. Dried blood spot analysis for therapeutic drug monitoring of pazopanib. J Clin Pharmacol. 2015 Dec;55(12):1344-50. doi: 10.1002/jcph.558. Epub 2015 Jul 14. PMID 26032288
- [Background] Nijenhuis CM, Huitema AD, Marchetti S, Blank C, Haanen JB, van Thienen JV, Rosing H, Schellens JH, Beijnen JH. The Use of Dried Blood Spots for Pharmacokinetic Monitoring of Vemurafenib Treatment in Melanoma Patients. J Clin Pharmacol. 2016 Oct;56(10):1307-12. doi: 10.1002/jcph.728. Epub 2016 Apr 8. PMID 26918324
- [Background] Ouellet D, Gibiansky E, Leonowens C, O'Hagan A, Haney P, Switzky J, Goodman VL. Population pharmacokinetics of dabrafenib, a BRAF inhibitor: effect of dose, time, covariates, and relationship with its metabolites. J Clin Pharmacol. 2014 Jun;54(6):696-706. doi: 10.1002/jcph.263. Epub 2014 Jan 17. PMID 24408395
- [Background] Friedl B, Kurlbaum M, Kroiss M, Fassnacht M, Scherf-Clavel O. A method for the minimally invasive drug monitoring of mitotane by means of volumetric absorptive microsampling for a home-based therapeutic drug monitoring. Anal Bioanal Chem. 2019 Jul;411(17):3951-3962. doi: 10.1007/s00216-019-01868-1. Epub 2019 May 16. PMID 31093700